CLINICAL TRIAL: NCT03681652
Title: Post-Operative Crohn's Disease Outcome in Children (The POPCORN Trial): a Prospective Comparative Non-interventional Open Study
Brief Title: Post-Operative Crohn's Disease Outcome in Children
Acronym: POPCORN
Status: Recruiting | Type: Observational
Sponsor: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Amit Assa, Head of IBD program, Schneider Children's Medical Center, Israel
Other Study IDs: POPCORN
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-11

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Azathioprine; Infliximab; CT-P13; Adalimumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Azathioprine or 6MP: Patients treated with thiopurines for post-operative prophylaxis.
  Interventions: Drug: Azathioprine
- Anti-TNF drug: Patients treated with anti-TNF alpha monotherapy for post-operative prophylaxis.
  Interventions: Drug: Anti-TNF Drug

INTERVENTIONS:
Drug: Azathioprine — Children with Crohn's disease who are treated with azathioprine for post-operative prophylaxis following ileo-cecal resection
  Other Names: Imuran
  Groups: Azathioprine or 6MP
Drug: Anti-TNF Drug — Children with Crohn's disease who are treated with anti-TNF monotherapy for post-operative prophylaxis following ileo-cecal resection
  Other Names: Remicade; Remsima; Humira
  Groups: Anti-TNF drug

SUMMARY:
Objectives: To examine the effect of prophylaxis therapy on clinical and endoscopic disease recurrence in children with Crohn's Disease (CD) following ileo-cecal resection. Hypothesis: Post-operative pediatric patients treated with anti-Tumor necrosis factor (TNF) prophylaxis will demonstrate lower endoscopic recurrence rates at 1 year and lower clinical recurrence rates at 2 years compared with thiopurines treated patients. Design: A multi-center, prospective, observational study. Patients with either thiopurines or anti-TNF prophylaxis will be enrolled 0-6 months following ileo-cecal resection. Prophylactic treatment will be decided at the discretion of the treating physician and not as a part of the study. According to standard-of-care, patients will undergo a colonoscopic evaluation 6-9 month following surgery. Study visits will be performed at 6 months following resection, 12 months, 18 months and 24 months. Setting: Porto group and IBD interest group pediatric gastroenterology centers. Participants: Children 6 year to 18 years (Overall, 84 patients) with CD following limited ileo-cecal resection. Main outcome measure: 1. Endoscopic recurrence at 1 year (according to Rutgeerts Score: i2-i4). 2. Clinical recurrence at 2 years (according to pediatric Crohn's disease activity index-PCDAI: ≥10). Secondary outcome measures: 1. Re-operation rate at 2 years. 2. Exacerbation-free quartiles at 2 years. 3. Anthropometric and laboratory measures including calprotectin at each visit. 4. Changes in fecal microbiome- baseline, 1 year and 2 years. Inclusion criteria: 1. CD with phenotypes L1 and L3 following ileo-cecal resection. 2. No active perianal disease. 3. Prophylactic therapy with either thiopurines or anti-TNF. Exclusion criteria: 1. Pregnancy. 2. Active perianal disease (draining fistula or abscess). 3. Post-operative intra-abdominal complication (fistula or abscess). Sample size: In order to demonstrate 20% difference in endoscopic recurrence rate between groups is significant, we will need to study 42 children in each group to be able to reject the null hypothesis that the failure rates between the groups are equal with probability (power) of 80% and a type I error probability of 0.05.

DETAILED DESCRIPTION:
Introduction Surgical intestinal resection of complicated or treatment refractory Crohn's disease (CD) is not uncommon. Ileocecal resection is the most frequent surgical intervention utilized in pediatric-onset CD, particularly in those with limited ileocecal disease. Only scarce data is available on the long-term outcome of patients following bowel resection in pediatric-onset CD . These studies have demonstrated that the risk for disease recurrence and additional surgical intervention is high in this population. Hence, as pediatric post-surgical patients are, by definition, high risk patients, prophylactic strategy is usually required. The most common prophylactic medications for post-operative recurrence are thiopurines and anti-TNF alpha agents. Adult randomized control trials assessing post-operative prophylaxis such as the PREVENT study and the POCER study have demonstrated similar short-term clinical recurrence rates (1 year) when comparing infliximab to placebo (PREVENT) or adalimumab to thiopurines (POCER). However, endoscopic recurrence rates did favor anti- tumor necrosis factor (TNF) prophylaxis. Apart from phenotypic characteristic and residual disease after resection there are data supporting fecal calprotectin as a strong predictor of disease recurrence. Both adult and pediatric guidelines recommend on performing a follow-up colonoscopy 6-9 month following surgical resection in-order to assess endoscopic activity by the Rutgeerts score and to adjust therapeutic regimens according to findings. Currently, there are no prospective or comparative studies assessing the effect of prophylactic post-operative therapies in children. Hence, it is the investigators aim is to assess the impact of postoperative prophylaxis on endoscopic and clinical recurrence in children with CD, following ileo-cecal resection using a prospective observational matched control design.

Hypothesis:

Post-operative pediatric patients treated with anti-TNF prophylaxis will demonstrate lower endoscopic recurrence rates at 1 year and lower clinical recurrence rates at 2 years compared with thiopurines treated patients.

Objectives:

Primary objective: To evaluate the effect of prophylactic therapy on clinical and endoscopic disease recurrence in children with CD following ileo-cecal resection.

Secondary objective: To evaluate the effect of prophylactic therapy on biochemical and anthropometric measures.

Methods:

Study design:

General design:

This is a multi-center, prospective, observational study with case-control matching. Patients with either thiopurines or anti-TNF alpha prophylaxis (including patients maintaining prior thiopurines and anti-TNF alpha treatment for post-operative prophylaxis) will be enrolled 0-3 months following ileo-cecal resection. Prophylactic treatment will be decided at the discretion of the treating physician and not as a part of the study. Medication regimen and dosage will be set by the treating physician according to standard of care and, agin, not as a part of the study. Patients will be enrolled at the first screening visit. Informed consent will be signed by both parents is required during enrollment. Informed assent will be offered for patients 14 years old and older. According to current recommended standard-of-care, patients will undergo a colonoscopic evaluation 6-9 month following surgery. Results will be documented according to the Rutgeerts score. Any other endoscopic or cross-sectional imaging performed during the study for clinical reasons will be documented in the appropriately.

Group 1: Patients treated with thiopurines for post-operative prophylaxis. Group 2: Patients treated with anti-TNF alpha monotherapy for post-operative prophylaxis.

Study Visits Scheduled visits will be performed at screening/enrolment (0-3 months following ileo-cecal resection) and at 6 months, 9 months, 12 months, 18 months and 24 months.

At enrollment, demographic, clinical, endoscopic, histologic and radiologic data will be retrieved, including with data on disease phenotype, course, therapeutic regimens, indication for surgery, type of surgery, surgical outcomes and pathology report from the resected specimen. Every visit all patients will be examined for height, weight, pediatric Crohn's disease activity index (PCDAI), physician global assesment (PGA) as well as comprehensive laboratory examinations including complete blood count (CBC), albumin, erythrocyte sedimentation rate (ESR) and C-reactive protein- CRP (CRP will be measured and registered in mg/dL). Fecal sample for fecal calprotectin will be obtained as well. At enrollment, 1 year and last visit fecal sample for microbiome analysis will be obtained.

Current treatment, and any treatment change since the previous visit will be recorded in the case report form. Relapse at any time should be noted along with PGA, and PCDAI at relapse.

Fecal calprotectin At each visit a single stool sample will be collected from each patient. One to 5 g stool will be stored at -20 degrees Celsius. Quantitative measurement of calprotectin will be performed using PhilCal Test (Calpro, Oslo, Norway) at the end of the study period at a central laboratory.

Fecal samples for microbiome Samples will be stored at -20ºc and then will be transported frozen to the laboratory where they were stored at -80ºc. Samples will be sent to a central laboratory at the end of the study (Sheba Medical Center, Tel Hashomer, Israel). DNA will be extracted from 200 mg of stool samples using Norgen Stool DNA extraction kit (Norgen Biotek) according to the manufacturer's instruction. The extracted DNA will be evaluated by agarose gel electrophoresis (1% w/v) and quantified spectrophotometrically. Libraries will be prepared and paired-end shotgun metagenomic sequencing will be performed on the Illumina MiSeq platform according to the manufacturer's specifications.

Anonymization and Coding Coding will be performed by the local principle investigator (PI) at enrollment according to site number and patient number. CRFs will not carry patients details apart from the code given by thr treating physician. Patients details can be identified and matched to the patient's code only by the local PI and for the purpose of filling missing data. Fecal Calprotectin tubes will be shifted using patients' codes only with no identified details.

Matching:

Patients will be matched between arms using case-control analysis according to baseline characteristics: Age, gender, indication for surgery, type of surgery, PCDAI following surgery, perianal disease, disease location/behavior, residual disease.

Data analysis:

Data will be analyzed using SPSS (version 25.0, SPSS, Inc., Chicago, IL, USA). Continuous variables will be evaluated for normal distribution using histogram, Q-Q Plots and Kolmogorov-Smirnov test and reported as median (interquartile range, IQR) for non-normally distributed variables or mean (standard deviation, SD) for normally distributed variables. Categorical variables will be reported as frequency and percentage. Continuous variables will be compared using independent simple T-test or Mann-Whitney while categorical variables will be compared using chi-square test or fisher-exact test. Correlation between continuous variables will be evaluated using Spearman rho correlation coefficient.

Patients with anti-TNF alpha prophylaxis will be matched to patients with thiopurines prophylaxis in a ratio of 1:1 (matched case-control). Patients will be matched as described earlier. Continuous variables will be compared between matched patients using paired sample T-test or Wilcoxon test while categorical variables will be compared using McNemar test. P-values <0.05 will be considered significant.

Sample size:

In order to demonstrate 20% difference in endoscopic recurrence rate between groups is significant, we will need to study 42 children in each group to be able to reject the null hypothesis that the failure rates between the groups are equal with probability (power) of 80% and a type I error probability of 0.05.

In-order to allow redundancy for non-matched patients, 50% non-matching rate is expected, thus requiring 100 patients.

Safety:

The study does not involve intervention. Any decision regarding prophylaxis initiation or treatment change during follow-up is at the sole discretion of the treating physician and not directed by the study. Clinical assessment is part of the routine follow-up of IBD patients. Blood samples are taken as standard of care along the course of the study with no extra blood samples needed. Colonoscopy at 6-9 months following ileo-cecal resection is considered standard of care and highly recommended by societal guidelines hence is not directed by the study but by accepted clinical guidelines. Nevertheless, a patient refusing colonoscopic evaluation as clinically indicated will remain in the study for the assessment of clinical recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Crohn's disease
2. Age: 6 - 17 years (inclusive)
3. L1 or L3 phenotypes
4. Ileocecal resection in the previous 3 months
5. No active perianal disease (including draining fistula or a peri-anal abscess)
6. Prophylactic therapy with either thiopurines or anti-TNF has been initiated

Exclusion Criteria:

1. Pregnancy
2. Renal Failure
3. Current abscess or perforation of the bowel
4. Post-operative intra-abdominal complication (fistula or abscess)
5. Complicated or heavily draining perianal fistula (indolent non-draining or minimally draining fistula are not an exclusion criteria).
6. Previous malignancy
7. Sepsis or active bacterial infection
8. IBD unclassified

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children at age 6 year to 17 years diagnosed with CD following first ileo-cecal resection.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Endoscopic recurrence (Rutgeerts score ≥ i2b) | 12 months following resection
  According to Rutgeerts score
  The Rutgeerts score:
  i0-no lesions in the neoterminal ileum i1-fewer than 5 aphthous lesions in the neoterminal ileum i2a-lesions confined to the ileocolonic anastomosis, including anastomotic stenosis), i2b-more than 5 aphthous ulcers or larger lesions, with normal mucosa in between, in the neoterminal ileum, with or without anastomotic lesions i3-diffuse aphthous ileitis with diffusely inflamed mucosa i4-large ulcers with diffuse mucosal inflammation or nodules or stenosis in the neoterminal ileum.

SECONDARY OUTCOMES:
Clinical recurrence according to PCDAI: ≥10 | 24 months
  According to PCDAI: ≥10
Re-operation rate | 24 months
  The rate of intra-abdominal re-operation
Exacerbation free quartiles | 24 months
  How many clinical flares were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Amit Assa, MD, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider Children's Hospital, Petah Tikva, Israel, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De Cruz P, Kamm MA, Hamilton AL, Ritchie KJ, Krejany EO, Gorelik A, Liew D, Prideaux L, Lawrance IC, Andrews JM, Bampton PA, Jakobovits S, Florin TH, Gibson PR, Debinski H, Gearry RB, Macrae FA, Leong RW, Kronborg I, Radford-Smith G, Selby W, Johnston MJ, Woods R, Elliott PR, Bell SJ, Brown SJ, Connell WR, Desmond PV. Efficacy of thiopurines and adalimumab in preventing Crohn's disease recurrence in high-risk patients - a POCER study analysis. Aliment Pharmacol Ther. 2015 Oct;42(7):867-79. doi: 10.1111/apt.13353. Epub 2015 Aug 28. PMID 26314275
- [Background] Rutgeerts P, Geboes K, Vantrappen G, Beyls J, Kerremans R, Hiele M. Predictability of the postoperative course of Crohn's disease. Gastroenterology. 1990 Oct;99(4):956-63. doi: 10.1016/0016-5085(90)90613-6. PMID 2394349